CLINICAL TRIAL: NCT03896542
Title: The Efficacy of Video Game Therapy in Patients With Stroke
Brief Title: The Effects of Video Games in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC 1559
Record Dates: First submitted 2019-03-15; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Commercial video game (Experimental): the group commercial video game received 30 minutes of conventional therapy plus 30 minutes of rehab training using Xbox Kinect-based games.
  Interventions: Device: Commercial video game.
- Rehabilitation video game (Experimental): the group rehabilitation video game received 30 minutes of conventional therapy plus 30 minutes of rehab games.
  Interventions: Device: rehabilitation video game
- The control group (No Intervention): The control group received 30 minutes of conventional therapy

INTERVENTIONS:
Device: Commercial video game. — Stroke patient had played with commercial video game, along 12 sessions.
  Arms: Commercial video game
Device: rehabilitation video game — Stroke patient had played with an specific video game for rehabilitation, along 12 sessions
  Arms: Rehabilitation video game

SUMMARY:
Aims: To establish whether the effectiveness of conventional treatment is increased when it is complemented with video-based therapy, whether specific rehabilitation or commercial after subacute stroke.

Design: Randomized clinical trial with pre / post-test and follow-up evaluation, assessor blinded study.

Methodology: Three different groups: conventional treatment, conventional treatment and commercial videogame, or conventional treatment and specific rehabilitation videogame. The three groups completed 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stroke
* Hemiplegia on the non-dominant side
* More than 1 month since the stroke
* Score 3 in the shoulder and 2 in the elbow in the modified Medical Research Council scale
* No auditory alterations
* No visual disturbances
* Mini Mental Scale greater than or equal to 24

Exclusion Criteria:

* Patients with unstable blood pressure or angina.
* History of seizures.
* Do not use video games

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Strength | Change from baseline at post 12 sessions of intervention and follow-up four weeks after having finished the intervention.
  The microFET 2© dynamometer had been used in order to evaluate the strength in several muscle groups: Shoulder (flexion and extension, adduction and abduction, internal and external rotation), elbow (flexion and extension, supination and pronation), wrist (flexion and extension).
Range of motion | Change from baseline at post 12 sessions of intervention and follow-up four weeks after having finished the intervention.
  The goniometer had been used in order to evaluate the range motion. Joints: Shoulder (flexion and extension, adduction and abduction, internal and external rotation), elbow (flexion and extension, supination and pronation), wrist (flexion and extension, ulnar and radial deviation ).

SECONDARY OUTCOMES:
Activities of daily living | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The Functional Independence Measure (FIM-FAM) measure was used to evaluate the independence in the activities of daily living
Fulg Meyer Assessment (FMA) | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The FMA was used to evaluated the upper limb function.
Box and Blocks test | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The Box and Blocks test was used to evaluate the manual dexterity in both upper limbs.
Muscle tone | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The Modified Ashworth scale has been used to evaluate the muscle tone. Muscle groups evaluated: Shoulder (flexion and extension, adduction and abduction, internal and external rotation), elbow (flexion and extension, supination and pronation), wrist (flexion and extension).

OTHER OUTCOMES:
The ID-Pain© the Lattineen Index. | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The ID-Pain was used to evaluate the pain.
Lattineen Index. | The measure was administrated in three times: pre intervention, post intervention (after 12 sessions carried out along four weeks) and follow-up four weeks after having finished the intervention.
  The Lattineen Index was used to evaluate the pain.

CONTACTS AND LOCATIONS:
Overall Officials: J. Hilario Ortiz Huerta, Principal Investigator — Universidad de Burgos
Locations (1):
- Universidad de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park DS, Lee DG, Lee K, Lee G. Effects of Virtual Reality Training using Xbox Kinect on Motor Function in Stroke Survivors: A Preliminary Study. J Stroke Cerebrovasc Dis. 2017 Oct;26(10):2313-2319. doi: 10.1016/j.jstrokecerebrovasdis.2017.05.019. Epub 2017 Jun 9. PMID 28606661
- [Background] Sin H, Lee G. Additional virtual reality training using Xbox Kinect in stroke survivors with hemiplegia. Am J Phys Med Rehabil. 2013 Oct;92(10):871-80. doi: 10.1097/PHM.0b013e3182a38e40. PMID 24051993
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2015 Feb 12;2015(2):CD008349. doi: 10.1002/14651858.CD008349.pub3. PMID 25927099
- [Background] Rand D, Weingarden H, Weiss R, Yacoby A, Reif S, Malka R, Shiller DA, Zeilig G. Self-training to improve UE function at the chronic stage post-stroke: a pilot randomized controlled trial. Disabil Rehabil. 2017 Jul;39(15):1541-1548. doi: 10.1080/09638288.2016.1239766. Epub 2016 Oct 28. PMID 27793071
- [Background] Gauthier LV, Kane C, Borstad A, Strahl N, Uswatte G, Taub E, Morris D, Hall A, Arakelian M, Mark V. Video Game Rehabilitation for Outpatient Stroke (VIGoROUS): protocol for a multi-center comparative effectiveness trial of in-home gamified constraint-induced movement therapy for rehabilitation of chronic upper extremity hemiparesis. BMC Neurol. 2017 Jun 8;17(1):109. doi: 10.1186/s12883-017-0888-0. PMID 28595611
- [Background] Bonnechere B, Jansen B, Omelina L, Van Sint Jan S. The use of commercial video games in rehabilitation: a systematic review. Int J Rehabil Res. 2016 Dec;39(4):277-290. doi: 10.1097/MRR.0000000000000190. PMID 27508968